CLINICAL TRIAL: NCT00001823
Title: Evaluation for NCI Surgery Branch Clinical Research Protocols
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990128; 99-C-0128; NCT00019799 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12-17

CONDITIONS: Synovial Cell Cancer; Melanoma; Colorectal Cancer; Lung Cancer; Bladder Cancer
Keywords: Cancer; Gene Therapy; Immunotherapy; Clinical Trial
MeSH Terms: conditions — Melanoma; Colorectal Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A/Surgery Branch Protocol Candidates: Patients suspected of having, or with biopsy proven, malignant disease being evaluated for or treated on NCI Surgery Branch protocols

SUMMARY:
Background:

The National Cancer Institute Surgery Branch (NCI-SB) has developed experimental therapies that involve taking white blood cells from patients' tumor or from their blood, growing them in the laboratory in large numbers, and then giving the cells back to the patient.

Objective:

This study will allow patients to under screening and evaluation for participation in NC-SB Protocols.

Eligibility:

Patients 18 years or older must meet the minimum eligibility criteria for an NCI-SB treatment protocol.

Design

Patients will undergo testing and evaluations as required by the appropriate NCI-SB treatment protocol.

DETAILED DESCRIPTION:
Background:

Potential research candidates undergo thorough screening including laboratory tests, scans, x-rays, and review of pathology slides to determine initial eligibility for National Cancer Institute Surgery Branch (NCI-SB) research protocols.

Objectives:

Permit evaluation of patients referred to the NCI-SB in order to identify individuals who will be suitable candidates for NCI-SB clinical research protocols.

To assess frequency of HLA type, gene specific mutations or expression of neo antigens in malignant tumors across the population of cancer patients undergoing screening for NCI-SB protocols.

Collect results of screening tests for use on subsequent research protocol as baseline (e.g., pretreatment) values.

Eligibility:

Age >= 18 years.

Patient suspected of having, or with biopsy proven, malignant disease.

Patient is able to understand and willing to sign a written informed consent document.

Patient is being evaluated for treatment on an NCI-SB protocols..

Design:

Patients enrolled on this protocol will be evaluated by NCI-SB physicians to determine the individual's suitability for participation in a clinical research protocol. An accrual ceiling of 7,000 patients has been set to meet the screening needs of the NCI-SB.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age >= 18 years.

Patient suspected of having, or with biopsy proven, malignant disease.

Patient is able to understand and willing to sign a written informed consent document.

Patient is being evaluated for treatment on an NCI-SB protocols.

EXCLUSION CRITERIA:

Women of child-bearing potential who are pregnant or plan to become pregnant because of the potentially dangerous effects of some of the screening procedures (e.g., nuclear medicine or other imaging scans) on the fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of having, or with biopsy proven, malignant disease.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 1999-07-11 (Actual)

PRIMARY OUTCOMES:
Number of individuals suitable for NCI Surgery Branch clinical research protocols | 25 Years
  Total number of patients who enroll on NCI Surgery Branch clinical research protocols
Frequency of HLA type, gene specific mutations, or expression of neoantigens in malignant tumors | 25 years
  Frequency of HLA type, gene specific mutations, or expression of neoantigens in tissue and blood samples
Results of screening tests | 25 years
  Results of screening tests for use on subsequent research protocol as baseline (e.g., pretreatment) values

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1999-C-0128.html